CLINICAL TRIAL: NCT02672020
Title: The COMETE Network, Towards an Easy-to-use Adrenal Cancer/Tumor Identity Card
Brief Title: Towards an Easy-to-use Adrenal Cancer/Tumor Identity Card
Acronym: COMETETACTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NI14028; PRTK-14-079 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2016-01-14; First posted 2016-02-03 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2016-01

CONDITIONS: Adrenal Gland Neoplasms
Keywords: pheochromocytoma; paraganglioma; adrenocortical carcinoma
MeSH Terms: conditions — Adrenal Gland Neoplasms; Pheochromocytoma; Paraganglioma; Adrenocortical Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with adrenal tumor (Experimental)
  Interventions: Biological: omics identity card

INTERVENTIONS:
Biological: omics identity card

SUMMARY:
Malignant pheochromocytoma/paraganglioma (MPP) and adrenocortical carcinoma (ACC) are two rare cancer entities with a very unfavorable prognosis. The knowledge on these rare cancers improved thanks to the French COMETE network originally based on two clinical centers (HEGP and Cochin) well organized for clinical and biological samples collection. Over the last 10 years, the COMETE key partners deciphered molecular mechanisms of tumorigenesis and oncogenesis of these tumors and identified molecular signatures discriminating between benign and malignant cancers by integrated genomic approaches. This strategy was highly successful in delivering new diagnostic applications of genomics technologies that now appear as potentially suitable for rapid implementation in routine clinical care.

The main objective of COMETE-TACTIC is to provide an easy-to-use "identity card" of the adrenal tumors that will allow a personalized "à la carte" management of the patient and, when indicated, to the indication of the most accurate molecular targeted therapy.

We hypothesize that the improvement of MPP and ACC diagnosis and of the therapeutic options proposed to affected patients will require,

1. the transfer to routine practice and the prospective validation of the novel diagnostic and predictive biomarkers issued from recent discoveries (genetics, genomics, histological biomarkers);
2. the implementation of the translational research projects based on the COMETE collection to identify circulating diagnostic, prognostic and therapeutic genetic and metabolic biomarkers that could be used as non-invasive "liquid biopsies".

DETAILED DESCRIPTION:
Malignant pheochromocytoma/paraganglioma (MPP) and adrenocortical carcinoma (ACC) are two rare cancer entities with a very unfavorable prognosis. The knowledge on these rare cancers improved thanks to the French COMETE ('COrtex, MEdulla Tumors Endocrines') network originally based on two clinical centers (HEGP and Cochin) well organized for clinical and biological samples collection. Over the last 10 years, the COMETE key partners deciphered molecular mechanisms of tumorigenesis and oncogenesis of these tumors and identified molecular signatures discriminating between benign and malignant cancers by integrated genomic approaches. COMETE has published more than 200 papers and performed seminal work on the pathophysiology and the genetics of MPP and ACC published in high-impact journals.

This strategy was highly successful in delivering new diagnostic applications of genomics technologies that now appear as potentially suitable for rapid implementation in routine clinical care.

The main objective of COMETE-TACTIC program is to design and validate an easy-to-use "identity card" classifying MPP and ACC in clinical routine, using molecular genomic and metabolomic tools combined with histopathological-based tests, to provide a real help for early diagnosis, prognostic as well as a personalized "à la carte" management and treatment to patients with malignant adrenal tumors. Seven teams, with an expertise in genomics of adrenal tumors, or in metabolomics approaches, or in clinical research and statistical analyses collaborate in COMETE-TACTIC. COMETE-TACTIC will be based on an already constituted large cohort of 850 patients that will be enlarged by the prospective enrolment of new cases and biological samples (300 to 450 new cases during the 3 years of the project) via 21 French expert and/or competence centers of COMETE-Cancer Reference center.

Previous COMETE basic studies provided important new insight for the understanding of molecular mechanisms responsible for MPP or ACC. With the transfer of "Omics"-based tests from research laboratories to clinical practice, COMETE-TACTIC is the next step toward a personalized medicine for patients with MPP and ACC. COMETE-TACTIC should speed the transfer in routine clinical care of new biomarkers based on cutting-edge technologies combining advanced pathology assessment and targeted genomics and metabolomics to diagnose malignancy and predict outcome, and thereby facilitating a more accurate, rapid and reliable diagnostic work-up for patients. This personalized management will help to avoid delayed diagnosis and to direct clinical decisions resulting in a better health outcome for the patients. COMETE-TACTIC will offer the access to a precise molecular classification of MPP and ACC that should guide targeted therapies. Finally, COMETE-TACTIC will investigate for the first time the impact of circulating biomarkers for the diagnosis and prognostic of adrenal cancers that will be further tested as biomarkers of response to targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated on a tumor developed from the adrenal cortex or a pheochromocytoma or a paraganglioma
* Age≥15 years
* Signature of the informed consent

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2015-11; Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Malignant status | Up to 36 months
  Number of participants with evidence of metastases

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Paule GIMENEZ-ROQUEPLO, Principal Investigator — Assistance Publique Hopitaux de Paris-HEGP, Paris, France
Locations (21):
- France (21):
  - CHU-Angers, Angers
  - CHU Rouen-Hopital de Bois-Guillaume, Bois-Guillaume
  - CHU Bordeaux, Hopital du Haut Leveque, Bordeaux
  - CHU Brest, Hopital de la Cavale Blanche, Brest
  - HCL- Centre Hospitalier Lyon Est, Bron
  - CHU Clermont-Ferrand, Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU Grenoble- Hopital Albert Michallon, Grenoble
  - Assistance Publique Hopitaux de Pais, Hopital de Bicetre, Le Kremlin-Bicêtre
  - CHU Limoges, Hopital du Cluzeau, Limoges
  - CHU Montpellier, Hopital Lapeyronie, Montpellier
  - CHU Nantes, Hopital Laënnec, Nantes
  - Assistance Publique Hopitaux de Paris -HEGP, Paris
  - Assistance Publique Hopitaux de Paris, Cochin, Paris
  - Assistance Publique Hopitaux de Paris, Necker, Paris
  - Assistance Publique Hopitaux de Paris, Pitie Salpetriere, Paris
  - CHU Reims, Hopital Robert Debre, Reims
  - CHU Rennes, Hopital Sud, Rennes
  - CHU Strasbourg, Hopital de Hautepierre, Strasbourg
  - CHU Toulouse, IUC Oncopole, Toulouse
  - CHU Tours, Hopital Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro-Vega LJ, Letouze E, Burnichon N, Buffet A, Disderot PH, Khalifa E, Loriot C, Elarouci N, Morin A, Menara M, Lepoutre-Lussey C, Badoual C, Sibony M, Dousset B, Libe R, Zinzindohoue F, Plouin PF, Bertherat J, Amar L, de Reynies A, Favier J, Gimenez-Roqueplo AP. Multi-omics analysis defines core genomic alterations in pheochromocytomas and paragangliomas. Nat Commun. 2015 Jan 27;6:6044. doi: 10.1038/ncomms7044. PMID 25625332
- [Background] Letouze E, Martinelli C, Loriot C, Burnichon N, Abermil N, Ottolenghi C, Janin M, Menara M, Nguyen AT, Benit P, Buffet A, Marcaillou C, Bertherat J, Amar L, Rustin P, De Reynies A, Gimenez-Roqueplo AP, Favier J. SDH mutations establish a hypermethylator phenotype in paraganglioma. Cancer Cell. 2013 Jun 10;23(6):739-52. doi: 10.1016/j.ccr.2013.04.018. Epub 2013 May 23. PMID 23707781
- [Background] Assie G, Letouze E, Fassnacht M, Jouinot A, Luscap W, Barreau O, Omeiri H, Rodriguez S, Perlemoine K, Rene-Corail F, Elarouci N, Sbiera S, Kroiss M, Allolio B, Waldmann J, Quinkler M, Mannelli M, Mantero F, Papathomas T, De Krijger R, Tabarin A, Kerlan V, Baudin E, Tissier F, Dousset B, Groussin L, Amar L, Clauser E, Bertagna X, Ragazzon B, Beuschlein F, Libe R, de Reynies A, Bertherat J. Integrated genomic characterization of adrenocortical carcinoma. Nat Genet. 2014 Jun;46(6):607-12. doi: 10.1038/ng.2953. Epub 2014 Apr 20. PMID 24747642